CLINICAL TRIAL: NCT05860309
Title: Preoperative Versus Postoperative Ultrasound Guided Quadratous Lunborum Block for Postoperative Analgesia Following Open Nephrectomy, Acomparative Study
Brief Title: Preoperative Versus Postoperative Quadratous Lunborum Block in Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sanaa Farag Mahmoud Wasfy, assistant professor of anesthesia and intensive care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS 183/2023
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Regional Blocks; Renal Surgery
Keywords: multimodal analgesia, regional blocks, renal surgeries

STUDY DESIGN:
Intervention Model Description: preoperative versus postoperative quadratous lumborum block in nephrectomy
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative quadratous lumborum block (Active Comparator): patients weill recieve preoperative ultrasound guided quadratous lumborum block at lateral position before start of surgery after induction of general anesthesia
  Interventions: Other: quadratous lumborum block
- postoperative quadratous lumborum block (Active Comparator): patients weill recieve postoperative ultrasound guided quadratous lumborum block at lateral position at the end of surgery before recovery from general anesthesua
  Interventions: Other: quadratous lumborum block

INTERVENTIONS:
Other: quadratous lumborum block — The patient will be placed in the lateral position, after sterilization.. QLB will be done using ultrasound, The probe will be positioned superior to the iliac crest, in the transverse orientation, at the posterior axillary line. The Shamrock sign will be identified at the L4 level, and the insulated nerve block needle will be advanced from posterior to anterior, through the QL muscle, until the needle tip is visualized in the interfascial plane between the QL muscle and psoas muscle. As the correct needle placement is confirmed with 2-3 mL of saline, 20 mL of 0.25% bupivacaine will be injected ensuring that the psoas muscle will be pushed deeply.
  Other Names: myofascial block

SUMMARY:
A multimodal analgesia regimen is suggested after nephrectomy, although some patients still report agonising pain. Regional anesthesia approaches may improve postoperative pain management and reduce the requirement for opioids after renal surgery.QLB provides early and rapid pain relief

DETAILED DESCRIPTION:
In the immediate postoperative period, nerve blocks are considered a type of multimodal analgesia and have recently been proposed as analgesic options for patients undergoing open nephrectomy .

Pain is defined as an unpleasant sensory and emotional experience associated with actual or potential tissue damage. The main barrier to early postoperative ambulation is postoperative pain, which also lengthens hospital stays and raises the risk of respiratory problems and venous thromboembolism. Therefore, strict perioperative pain management can have both immediate and long-term advantages .

QLB provides early and rapid pain relief and allows early ambulation in certain patient populations. Multiple case studies also confirmed the QLB to be a rescue block after different surgical procedures. Complications associated with the performance of abdominal wall blocks are fortunately very rare. However, studies on the effect of anterior QLB on postoperative opioid consumption are scarce .

Regional anesthesia is quickly moving toward using ultrasound guidance as the gold standard. The use of ultrasound has significant advantages over traditional treatments such as nerve stimulation and loss of resistance. The improved safety and efficacy that ultrasound brings to regional anaesthesia will help promote its use and realise the benefits that regional anaesthesia has over general anaesthesia, such as decreased morbidity and mortality, superior postoperative analgesia, cost-effectiveness, decreased postoperative complications and an improved postoperative course .

The aim of the present study is to compare the effectiveness of ultrasound-guided preoperative to postoperative QLB on the postoperative pain scores after Radical nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* o Patients aged between 18 - 60 years old.

  * Both sexes.
  * Physical Status: ASA I and II.

Exclusion Criteria:

* o Refusal of procedure or participation in the study .

  * Physical status: ASA III or above .
  * Infection at site of injection.
  * Psychiatric illness .
  * CNS Diseases like epilepsy, stroke …etc.
  * History or evidence of coagulopathy .
  * Allergies to drug used (Bupivacaine 0.5%).
  * Patients who suffered from allergy to local anesthetics .
  * Difficult visualization of the anatomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The time to first postoperative rescue analgesia. | postoperative 24 hours
  the first time patient ask for analgesia

SECONDARY OUTCOMES:
total consumption of opioid in first 24 hours | first 24 hours postoperatively
  amount of narcotic needed by patient in first 24 hours after nephrectomy

CONTACTS AND LOCATIONS:
Overall Officials: sanaa F wasfy, Principal Investigator — Ain Shams University
Locations (1):
- Ainshams hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borys M, Szajowska P, Jednakiewicz M, Wita G, Czarnik T, Mieszkowski M, Tuyakov B, Galkin P, Rahnama-Hezavah M, Czuczwar M, Piwowarczyk P. Quadratus Lumborum Block Reduces Postoperative Opioid Consumption and Decreases Persistent Postoperative Pain Severity in Patients Undergoing Both Open and Laparoscopic Nephrectomies-A Randomized Controlled Trial. J Clin Med. 2021 Aug 15;10(16):3590. doi: 10.3390/jcm10163590. PMID 34441884